CLINICAL TRIAL: NCT02038101
Title: Feedback and Education Intervention to Reduce Inappropriate Transthoracic Echocardiograms (TTE)
Brief Title: A Multi-centered Feedback and Education Intervention Designed to Reduce Inappropriate Transthoracic Echocardiograms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other); Scarborough General Hospital (Other); Kingston Health Sciences Centre (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WCHTTE-001
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: CARDIOVASCULAR DISEASES
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and Feedback Intervention (Experimental): This intervention includes the following components:
  1. Formal Rounds on AUC for TTE:
  2. Appropriate Use for TTE Application for Smartphone
  3. Individualized Feedback Reports provided by email
  Interventions: Behavioral: Education and Feedback
- Control (No Intervention): Usual echocardiography ordering pratice.

INTERVENTIONS:
Behavioral: Education and Feedback — 1. Formal Rounds on AUC for TTE
  2. Appropriate Use for TTE Application for Smartphone
  3. Individualized Feedback Reports provided by email
  Arms: Education and Feedback Intervention

SUMMARY:
This study is an international, prospective, multi-centred, investigator blinded, randomized control trial of an educational and feedback-based intervention vs. usual care to study the proportion of inappropriate TTEs ordered by clinicians in ambulatory care.

The American College of Cardiology collaborated with the American Society of Echocardiography to develop its Appropriate Use Criteria (AUC) for Echocardiography in 2007, and were updated in 2011.

We created an innovative education and feedback-based intervention that we hypothesize will reduce the proportion of inappropriate TTEs ordered in clinical practice. Our objective is to prospectively study the following intervention in a multicentre, randomized control trial format to determine if this intervention will reduce inappropriate TTEs and the number of TTEs ordered in practice.

The study will take place at multiple hospitals in Canada the United States. Participants include cardiologists and primary care providers (both general internal medicine and family practice) who provide ambulatory care.

Once cardiologists and primary care physicians are recruited for the study, they will be randomized into one of two arms: 1) Intervention group, 2) Control group.

A physician's TTE ordering information will be ascertained by review of the individual TTE order and by review of the patient's medical record. Trained research coordinators at each site will review the TTE order for indication and review the patient record to ascertain clinical circumstances regarding the TTE order. The individual research coordinator will review this information using the 2011 AUC and classify the TTE as Appropriate (A), Inappropriate (I) or Uncertain (U), and assign the TTE order the most appropriate indication number accordingly. Research Coordinators will be blinded to which physicians are in the intervention or control group.

Research Coordinators at each site will be responsible for individual physicians' TTE order classifications but will be blinded to study group. Once monthly TTE orders are classified and collated, this information will be transmitted to the central research laboratory, where a research coordinator will collate all of the results and transmit monthly feedback reports to individual physicians. The control group will order TTEs as is their usual practice.

DETAILED DESCRIPTION:
This study is an international, prospective, multi-centred, investigator blinded, randomized control trial of an educational and feedback-based intervention vs. usual care to study the proportion of inappropriate TTEs ordered by clinicians in ambulatory care.

Increased inappropriate TTE utilization represents a burden to health budgets as costs rise with increased utilization, and to patients themselves who are burdened with unnecessary procedures that can adversely affect quality of care. Rising utilization in an environment with limited supply also creates barriers to access and increased wait times for those patients in the community who are awaiting necessary TTEs.

In a move to balance the concern regarding rising utilization while still ensuring physician autonomy on access to ordering cardiac tests and procedures, the American College of Cardiology collaborated with the American Society of Echocardiography to develop its Appropriate Use Criteria (AUC) for Echocardiography in 2007, and were updated in 2011. AUC were created by using the modified RAND appropriateness method. Studies applying AUC to TTE orders at single centres in the US found inappropriate TTE rates in ambulatory (outpatient) care ranging up to 35%.

We have successfully created an innovative education and feedback-based intervention that we hypothesize will reduce the proportion of inappropriate TTEs ordered in clinical practice, which will save healthcare dollars and improve quality of care and access to echocardiography. Our objective is to prospectively study the following intervention in a multicentre, randomized control trial format to determine if this intervention will reduce inappropriate TTEs and the number of TTEs ordered in practice.

The study will take place at multiple hospitals in Canada the United States. Participants include cardiologists and primary care providers (both general internal medicine and family practice) who provide ambulatory care. Only providers who see patients in ambulatory care clinics will be included. Pediatric cardiologists and physicians who specialize primarily in adult congenital heart disease will be excluded from the study. Physicians who are approached will be required to provide written consent prior to participation in the study.

Once cardiologists and primary care physicians are recruited for the study, they will be randomized into one of two arms: 1) Intervention group, 2) Control group. Randomization will occur at the same time for each site to ensure the study start date is consistent across all sites.

Collection of TTE ordering information and TTE order classification:

A physician's TTE ordering information will be ascertained by review of the individual TTE order and by review of the patient's medical record. This may be through review of the Electronic Medical Record (EMR) or paper chart, depending on the individual site. Trained research coordinators at each site will review the TTE order for indication and review the patient record to ascertain clinical circumstances regarding the TTE order. The individual research coordinator will review this information using the 2011 AUC and classify the TTE as Appropriate (A), Inappropriate (I) or Uncertain (U), and assign the TTE order the most appropriate indication number accordingly. TTE orders that do not have a corresponding indication number will be designated as unclassifiable. Research Coordinators will be blinded to which physicians are in the intervention or control group. This system of TTE classification has been previously piloted and published by our group in two recently published studies, and the rate of successful classification was greater than 98%.

Dissemination of TTE monthly feedback reports:

Research Coordinators at each site will be responsible for individual physicians' TTE order classifications but will be blinded to study group. Once monthly TTE orders are classified and collated, this information will be transmitted to the central research laboratory, where a research coordinator will collate all of the results and transmit monthly feedback reports to individual physicians. This process ensures that local site coordinators and the study investigators are blinded to the results to the study, while still enabling the creation and dissemination of physician related feedback reports to the intervention group. The control group will order TTEs as is their usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Cardiologist or physician practicing Primary Care in the Ambulatory care

Exclusion Criteria:

* . Pediatric cardiologists and physicians who specialize primarily in adult congenital heart disease will be excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of Inappropriate Transthoracic Echocardiograms ordered (%) | 18 months

SECONDARY OUTCOMES:
Total Number of Transthoracic Echocardiograms Ordered per Physician | 18 months

OTHER OUTCOMES:
Proportion of Appropriate Transthoracic Echocardiograms Ordered (%) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sacha R Bhatia, MD, Principal Investigator — Women's College Hospital
Locations (6):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in an academic peer-reviewed journal.

REFERENCES:
- [Background] Bhatia RS, Milford CE, Picard MH, Weiner RB. An educational intervention reduces the rate of inappropriate echocardiograms on an inpatient medical service. JACC Cardiovasc Imaging. 2013 May;6(5):545-55. doi: 10.1016/j.jcmg.2013.01.010. Epub 2013 Apr 10. PMID 23582360
- [Background] Blecker S, Bhatia RS, You JJ, Lee DS, Alter DA, Wang JT, Wong HJ, Tu JV. Temporal trends in the utilization of echocardiography in Ontario, 2001 to 2009. JACC Cardiovasc Imaging. 2013 Apr;6(4):515-22. doi: 10.1016/j.jcmg.2012.10.026. PMID 23579013
- [Background] Bhatia RS, Carne DM, Picard MH, Weiner RB. Comparison of the 2007 and 2011 appropriate use criteria for transthoracic echocardiography in various clinical settings. J Am Soc Echocardiogr. 2012 Nov;25(11):1162-9. doi: 10.1016/j.echo.2012.07.018. Epub 2012 Aug 14. PMID 22898245
- [Derived] Tharmaratnam T, Bouck Z, Sivaswamy A, Wijeysundera HC, Chu C, Yin CX, Nesbitt GC, Edwards J, Yared K, Wong B, Weinerman A, Thavendiranathan P, Rakowski H, Dorian P, Anderson G, Austin PC, Dudzinski DM, Ko DT, Weiner RB, Bhatia RS. Association Between Physicians' Appropriate Use of Echocardiography and Subsequent Healthcare Use and Outcomes in Patients With Heart Failure. J Am Heart Assoc. 2020 Jan 7;9(1):e013360. doi: 10.1161/JAHA.119.013360. Epub 2019 Dec 24. PMID 31870231
- [Derived] Tharmaratnam T, Bouck Z, Sivaswamy A, Wijeysundera HC, Chu C, Yin CX, Nesbitt GC, Edwards J, Yared K, Wong B, Weinerman A, Thavendiranathan P, Rakowski H, Dorian P, Anderson G, Austin PC, Dudzinski DM, Ko DT, Weiner RB, Bhatia RS. Low-Value Transthoracic Echocardiography, Healthcare Utilization, and Clinical Outcomes in Patients With Coronary Artery Disease. Circ Cardiovasc Qual Outcomes. 2019 Nov;12(11):e006123. doi: 10.1161/CIRCOUTCOMES.119.006123. Epub 2019 Nov 11. PMID 31707824
- [Derived] Bhatia RS, Ivers NM, Yin XC, Myers D, Nesbitt GC, Edwards J, Yared K, Wadhera RK, Wu JC, Kithcart AP, Wong BM, Hansen MS, Weinerman AS, Shadowitz S, Elman D, Farkouh ME, Thavendiranathan P, Udell JA, Johri AM, Chow CM, Hall J, Bouck Z, Cohen A, Thorpe KE, Rakowski H, Picard MH, Weiner RB. Improving the Appropriate Use of Transthoracic Echocardiography: The Echo WISELY Trial. J Am Coll Cardiol. 2017 Aug 29;70(9):1135-1144. doi: 10.1016/j.jacc.2017.06.065. PMID 28838362
- [Derived] Bhatia RS, Ivers N, Yin CX, Myers D, Nesbitt G, Edwards J, Yared K, Wadhera R, Wu JC, Wong B, Hansen M, Weinerman A, Shadowitz S, Johri A, Farkouh M, Thavendiranathan P, Udell JA, Rambihar S, Chow CM, Hall J, Thorpe KE, Rakowski H, Weiner RB. Design and methods of the Echo WISELY (Will Inappropriate Scenarios for Echocardiography Lessen SignificantlY) study: An investigator-blinded randomized controlled trial of education and feedback intervention to reduce inappropriate echocardiograms. Am Heart J. 2015 Aug;170(2):202-9. doi: 10.1016/j.ahj.2015.04.022. Epub 2015 May 1. PMID 26299215